CLINICAL TRIAL: NCT01152125
Title: Use of Autologous Bone Marrow Stem Cell Transplantation for Therapeutic Chondrogenesis in Moderate to Severe Osteoarthritis - ABM & LAM ST-OA Study
Brief Title: Safety and Efficacy of Autologous Bone Marrow Stem Cells for Treating Osteoarthritis
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: International Stemcell Services Limited (Industry)
Responsible Party: Dr. SGA Rao, Chairman, International Stemcell Services Ltd.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ISSL-AuBM-OA
Record Dates: First submitted 2010-06-25; First posted 2010-06-29 (Estimated); Last update posted 2011-06-09 (Estimated); Status verified 2011-06

CONDITIONS: Osteoarthritis
Keywords: Osteoarthritis; stem cell implantation; bone marrow; autologous
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Autologous bone marrow stem cells (Experimental)
  Interventions: Other: Autologous bone marrow stem cells

INTERVENTIONS:
Other: Autologous bone marrow stem cells — Stem cells isolated from the patient's own bone marrow.

SUMMARY:
Osteoarthritis is a leading cause of chronic disability in elderly and the risk of disability attributed to osteoarthritis is as great as or greater than due to any other medical condition in that age group. Several cross sectional studies have demonstrated an age related increase in the prevalence of osteoarthritis of knee(5). Results of survey are similar with most surgeons reporting 50+ years age group being commonest at initial presentation and that the incidence increases with advancing age. Interestingly some surgeons have noticed earlier occurrence of osteoarthritis in 40+ years age group and one has to be careful to screen for secondary causes in this younger age group patients.

While pain relief is the primary treatment goal of osteoarthritis medications, localized inflammation may also be relieved by using certain drugs. Managing osteoarthritis pain can involve medications, natural remedies, exercise, weight loss, joint protection, mobility aids, assisted devices and more.

Stem cell therapy, using cells extracted from the same patient or suitable alternative human sources, targets diseases which are either incurable or with no complete or effective treatment available in the traditional healthcare system. Since this therapy is based on the concept of regenerating damaged cells in the injured or disease-affected areas of the body, it is called regenerative medicine

Autologous stem cells provide an attractive option for osteoarthritis patients and their clinicians.

In our present study we want to evaluate the safety and efficacy of autologous bone marrow derived stem cells in treatment of Osteoarthritis for therapeutic chondrogenesis through delivery of stem cells into the knee joint space in ten Indian patients.

ELIGIBILITY:
Inclusion Criteria:

1. Must be able to give voluntary written (patients may not be able to write) consent.
2. Must be able to understand study information provided to him.
3. Age 30 to 70, inclusive
4. OA Kellgren and Lawrence classification 3 & 4
5. No ligamentous laxity i.e. stable
6. Ability to understand and willingness to sign consent form
7. The participant is able to comply with and understand the required visit schedule and all required tests and procedures.

Exclusion Criteria:

1. Serious pre-existing medical conditions like Diabetes Mellitus, Chronic Renal Failure, Rheumatoid Arthritis, Collagen vascular diseases and Autoimmune diseases
2. Pregnant or lactating woman
3. Inflammatory arthritis
4. Oral steroid, methotrexate (immune suppressants)
5. History of drug or alcohol abuse or chronic smoking
6. Poor patient compliance
7. Infectious disease test positive for HIV 1&2, HbsAg, HCV and VDRL.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2010-01; Primary Completion 2011-08 (Estimated); Study Completion 2012-01 (Estimated)

PRIMARY OUTCOMES:
Pain as measured by the The Western Ontario and McMaster Universities Arthritis Index (WOMAC) Pain Score | Baseline, 3 months, 6 months, 1 year
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 1 year

SECONDARY OUTCOMES:
Changes in the MRI knee with cartilage mapping and clinical improvement | Baseline, 6 months, 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Rudraprasad, M.S, Principal Investigator — St. Theresa's Hospital; Alphy Zachson, M.B.B.S, Study Director — International Stemcell Services Limited
Locations (1):
- St. Theresa's Hospital, Bengaluru, Karnataka, India